CLINICAL TRIAL: NCT05504161
Title: Detection of Tumor DNA Through Cervical Smear and Liquid Biopsy in Endometrial Cancer Patients and Evaluation of Prognostic and Predictive Values of Tumor DNA Assay
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2020-1265
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor genomic DNA from cervical swab and cell-free DNA from frozen plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endometrial cancer group: Patients pathologically diagnosed with endometrial cancer
- Control group: Patients with benign endometrial pathology and interepithelial neoplasia

SUMMARY:
Circulating tumor DNA (ctDNA) may help detect and prognosis-stratify patients with endometrial cancer. Both cervical swab-based genomic DNA (gDNA) and whole blood-based ctDNA can be utilized for this goal. Our objective is to utilize cervical swab and whole blood samples to analyze tumor-derived ctDNA from patients with endometrial cancer. These samples will be collected prospectively, and prior to staging operation. Samples from patients without cancer, who undergo hysterectomy for benign gynecological cause, will be utilized as controls. Variants called by next generation sequencing were classified into four-tiers based on ASCO/AMP system. These initially captured samples will be used to compare performance in terms of detection rate and to stratify patients based on the mutational profile. Additionally, in patients with advanced disease, we plan to collect whole blood samples every 3 months to assess any changes in mutational landscape. Clinical data including age, cormorbidities, treatment methods, date of diagnosis and recurrence, response evaluation for chemotherapy or radiotherapy, survival data will be used to contextualize our findings.

ELIGIBILITY:
Inclusion Criteria:

1. Female, over 19 years of age
2. Patients with endometrial cancer or benign gynecological diseases

Exclusion Criteria:

1. Patients in pregnancy
2. Patients being treated for cancer of other organs, including gynecological cancer.
3. Patients who has difficulty reading and understanding Korean.
4. The tester's determination that the patient will not be able to comply with the clinical trial procedures.
5. Patients with severe infections or other serious medical problems that have resulted in impairment of the patient's function, making it difficult to the trial.

Ages: 19 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are diagnosed endometrial cancer (case) and benign gynecological disease (control)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-12-30 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Detection rate | Detection rate based on two different modalities at the time of surgery.
  We aim to compare the ctDNA mutation detection rate based on cervical swab and whole blood at the time of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Yun Lee, M.D., Principal Investigator — Department of Obstetrics and Gynecology, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No